CLINICAL TRIAL: NCT00494065
Title: Chiropractic and Self-care for Back-Related Leg Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern Health Sciences University (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18HP07638; R18HP07638
Record Dates: First submitted 2007-06-27; First posted 2007-06-29 (Estimated); Last update posted 2014-01-31 (Estimated); Status verified 2014-01

CONDITIONS: Sub-acute and Chronic Back-related Leg Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- 1 (Experimental): Chiropractic Spinal Manipulative Therapy + Home exercise
  Interventions: Other: Chiropractic Spinal Manipulative Therapy + Home exercise
- 2 (Active Comparator): Home exercise
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Home exercise — Patient education will be provided by trained therapists under the supervision of licensed chiropractic clinicians. Patients will attend four, 1 hour, one-on-one sessions.
  Arms: 2
Other: Chiropractic Spinal Manipulative Therapy + Home exercise — The number and frequency of treatments will be determined by the individual chiropractor, based on patient-rated symptoms, disability, palpation, and pain provocation tests. Up to 20 treatments will be provided over the 12 week treatment period, each treatment visit lasting from 10-20 minutes. Treatment will include manual spinal manipulation and mobilization.
  Arms: 1

SUMMARY:
The primary aims of the project are to determine the clinical efficacy of chiropractic Spinal Manipulative Therapy (SMT) plus self-care education versus self-care education alone in 192 patients with sub-acute and chronic Back Related Leg Pain (BRLP) in both the short-term (after 12 weeks) and long-term (after 52 weeks). The primary outcome variable is leg pain and secondary outcome variables include low back pain, disability, bothersomeness and frequency of symptoms, general health status, and fear avoidance behavior.

Secondary aims are to describe and estimate between group differences in patient satisfaction, improvement, medication use, straight leg raise, torso endurance, and three biomechanical measures: continuous spinal motion, postural sway, and neuromuscular response to sudden load. Patient perceptions of treatment will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Back-related leg pain > 3 on 0 to 10 scale.
* Sub-acute or chronic back-related leg pain defined as current episode > 4 weeks duration.
* Back-related leg pain classified as 2, 3, 4, or 6 using the Quebec Task Force (QTF) Classification system. This includes radiating pain into the proximal or distal part of the lower extremity, with or without neurological signs, with possible compression of a nerve root.
* 21 years of age and older.
* Stable prescription medication plan (no changes in prescription medications that affect musculoskeletal pain in the previous month).

Exclusion Criteria:

* Ongoing treatment for leg or low back pain by other health care providers.
* Progressive neurological deficits or cauda equina syndrome.
* QTF classifications 5 (spinal fracture) and 11 (other diagnoses including visceral diseases, compression fractures, metastases). These are serious conditions not amenable to the conservative treatments proposed.
* QTF 7 (spinal stenosis syndrome characterized by pain and/or paresthesias in one or both legs aggravated by walking).
* Uncontrolled hypertension or metabolic disease.
* Blood clotting disorders.
* Severe osteoporosis.
* Inflammatory or destructive tissue changes of the spine.
* Patients with surgical lumbar spine fusion or patients with multiple incidents of lumbar surgery. This is a subgroup of low back pain patients which generally have a poorer prognosis.
* Pregnant or nursing women.
* Current or pending litigation. Patients seeking financial compensation tend to respond differently to treatment.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2007-06; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Patient-rated leg pain | short-term = 12 weeks; long-term = 52 weeks

SECONDARY OUTCOMES:
Bothersomeness | short-term = 12 weeks; long-term = 52 weeks
Frequency | short-term = 12 weeks; long-term = 52 weeks
Disability | short-term = 12 weeks; long-term = 52 weeks
General Health Status | short-term = 12 weeks; long-term = 52 weeks
Fear Avoidance | short-term = 12 weeks; long-term = 52 weeks
Patient Satisfaction | short-term = 12 weeks; long-term = 52 weeks
Improvement | short-term = 12 weeks; long-term = 52 weeks
Medication Use | short-term = 12 weeks; long-term = 52 weeks
Biomechanical test measures: Continuous lumbar motion, Standing postural sway, Neuromuscular response to a sudden load, Straight leg raise test, Torso muscle endurance | short-term = 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gert Bronfort, DC, PhD, Principal Investigator — Northwestern Health Sciences University
Locations (2):
- United States (2):
  - Palmer Center for Chiropractic Research, Davenport, Iowa
  - Northwestern Health Sciences University, Bloomington, Minnesota

REFERENCES:
- [Derived] Bronfort G, Hondras MA, Schulz CA, Evans RL, Long CR, Grimm R. Spinal manipulation and home exercise with advice for subacute and chronic back-related leg pain: a trial with adaptive allocation. Ann Intern Med. 2014 Sep 16;161(6):381-91. doi: 10.7326/M14-0006. PMID 25222385
- [Derived] Schulz CA, Hondras MA, Evans RL, Gudavalli MR, Long CR, Owens EF, Wilder DG, Bronfort G. Chiropractic and self-care for back-related leg pain: design of a randomized clinical trial. Chiropr Man Therap. 2011 Mar 22;19:8. doi: 10.1186/2045-709X-19-8. PMID 21426558